CLINICAL TRIAL: NCT00435916
Title: A Phase II Study of SGN-40 (Anti-huCD40 mAb) in Patients With Relapsed Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Study of SGN-40 in Patients With Relapsed Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG040-0004
Record Dates: First submitted 2007-02-14; First posted 2007-02-16 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin
Keywords: Antigens, CD40; Antibody, Monoclonal; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Lymphoma | interventions — dacetuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SGN-40

INTERVENTIONS:
Drug: SGN-40 — 1-8 mg/kg IV (in the vein) on Days 1, 4, 8, 15, 22 and 29 of Cycle 1; 8 mg/kg IV (in the vein) on Days 1, 8, 15, and 22 for Cycles 2-12.
  Other Names: dacetuzumab

SUMMARY:
This is a Phase II, open-label, multidose trial of SGN-40 designed to estimate objective response rate and assess toxicity in patients with relapsed DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DLBCL.
* Received at least one combination chemotherapy regimen with rituximab, such as R-CHOP, R-ESHAP or equivalent.
* Progression or relapse since most recent therapy.
* At least one measurable lesion that is both greater than or equal to 2 cm by conventional CT or greater than or equal to 1.5 cm by spiral CT.

Exclusion Criteria:

* Previous diagnosis or treatment for indolent lymphoma, leptomeningeal lymphoma, or central nervous system lymphoma.
* Primary refractory disease.
* Received an allogenic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Objective response as assessed by CT and PET scans and revised response criteria for malignant lymphoma. | Every 1 or 2 months

SECONDARY OUTCOMES:
Progression-free survival, disease-free survival, and overall survival. | Study duration
Adverse events, laboratory values, and anti-drug antibody immune responses. | Within 3 weeks of final infusion
PK profile. | Within 3 weeks of final infusion

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Whiting, PharmD, Study Director — Seagen Inc.
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic-Arizona, Scottsdale, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Sharp Healthcare, San Diego, California
  - Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Swedish Cancer Institute, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] de Vos S, Forero-Torres A, Ansell SM, Kahl B, Cheson BD, Bartlett NL, Furman RR, Winter JN, Kaplan H, Timmerman J, Whiting NC, Drachman JG, Advani R. A phase II study of dacetuzumab (SGN-40) in patients with relapsed diffuse large B-cell lymphoma (DLBCL) and correlative analyses of patient-specific factors. J Hematol Oncol. 2014 Jun 12;7:44. doi: 10.1186/1756-8722-7-44. PMID 24919462